CLINICAL TRIAL: NCT07313592
Title: A Prospective Study of Whole Genome Sequencing (ChromoSeq®) at Diagnosis for Pediatric, Adolescent, and Young Adult Acute Lymphoblastic Leukemia (ALL) Patients
Brief Title: Whole Genome Sequencing (ChromoSeq®) for Acute Lymphoblastic Leukemia (ALL) Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: McDonnell Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202512057
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; B-ALL; T-ALL; Next generation sequencing; Pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow aspirate specimen and/or 1 mL of peripheral blood collection will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Child and Young Adult acute lymphoid leukemia (ALL) patients: At time of initial workup, patients will undergo bone marrow and/or peripheral blood collection for ChromoSeq® (requires 1 mL of peripheral blood or bone marrow aspirate).
  Interventions: Device: ChromoSeq® assay testing

INTERVENTIONS:
Device: ChromoSeq® assay testing — Bone marrow and/or peripheral blood sample will be collected and ChromoSeq® assay testing will be completed.

SUMMARY:
This is a prospective specimen collection study evaluating the feasibility of using the ChromoSeq® assay for upfront classification in a real-time clinical setting of pediatric and young adult acute lymphoid leukemia (ALL) patients. Sixty patients will undergo collections of bone marrow and/or peripheral blood for the ChromoSeq® assay at time of initial workup, and the patients will then be followed for clinical outcomes for up to 65 months.

ELIGIBILITY:
Eligibility Criteria

* Children and young adult patients (< 30 years of age at time of study enrollment) treated at St. Louis Children's Hospital/Washington University School of Medicine.
* Suspected diagnosis or suspected relapse of acute lymphoblastic leukemia (ALL), B- or T-cell.
* Concurrent enrollment on a prospective therapeutic trial is allowed as this protocol makes no recommendations regarding treatment approach.
* Ability to understand and willingness to sign an IRB approved written informed consent document. All patients and/or their parents or legal guardians must sign an IRB approved written informed consent document.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Child and young adult patients diagnosed with acute lymphoid leukemia (ALL) seen at St. Louis Children's Hospital/Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Rate of success of ChromoSeq® | Time of specimen collection to completion of results (total estimated time is 15 days)
  ChromoSeq® will be successful if the results on the first attempt in a real-time, clinical setting identifies recurrent structural variants and copy number alterations of conventional cytogenetics and karyotype. The success rate and the 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Comparison of time-to-results of ChromoSeq® and conventional cytogenetics | Time of specimen collection to 15 days after collection (total estimated time is 15 days)
  The proportion of results return within 15 days and the 95% confidence interval will be calculated.
Frequency of mismatch between LDA standard testing and ChromoSeq® defined Ph-like patients. | Time of specimen collection to completion of LDA testing (total estimated time is 15 days)
  The outcome will be measured by determining the correlation of LDA testing on patients with neutral cytogenetics versus LDA testing on patients whose ChromoSeq® results display a Ph-like translocation for validation.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Ferris, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be uploaded to dbGaP.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu